CLINICAL TRIAL: NCT04393857
Title: The Temporo-spatial Dynamics of Genital Tract Microbiota - an Observational Study in Oocyte Donors
Status: Completed | Type: Observational
Sponsor: Peter Humaidan (Other)
Collaborators: Instituto Bernabeu (Other)
Responsible Party: Sponsor-Investigator, Peter Humaidan, Professor, Consultant, Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Other Study IDs: Microbiome_endometrial_spain
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Bacterial Vaginoses
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Vaginal, Cervical and endometrial samples taken with the Eswab (Copan), eNAT (Copan) and Tao brush (Cook medical). Although there will be Human DNA in samples, we aim to isolate bacterial DNA for further analysis. No analyses are planned on Human DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oocyte donors: Healthy Oocyte donors fulfilling the criteria for oocyte donation are eligible. Patients may not have received any antibiotics or vaginal products (other than for menstrual hygiene - such as tampons) for the last 1 month. Informed consent is mandatory.

SUMMARY:
The investigators aim to examine the endometrium with state of the art sequencing techniques to investigate the endometrial microbiota. The endometrial microbiota has been perceived to be sterile, however, this seems incorrect from recent studies. Thus, the primary outcome is to compare the rate of ascending infection from the vagina to the endometrium and to investigate which bacteria are capable of inhabiting these environments in healthy oocyte donors. These results will be compared to equivalent samples of IVF patients.

ELIGIBILITY:
Inclusion Criteria:

Oocyte donors meeting local criteria for donation. Written informed consent. Regular cycle

Exclusion Criteria:

Antibiotics within 1 month Vaginal products other than for menstrual hygiene within 1 month Uterine malformations(Septum, polyps, adenomyosis, fibroids) HIV, Hepatitis B or C positivity. HPV CIN 2 or higher. Chlamydia trachomatis positivity.

Any uncontrolled concomitant disease (e.g. uncontrolled diabetes, uncontrolled hypertension etc.)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy oocyte donors
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of ascending infection/sharing of bacteria in the genital tract | This outcome data is measured at the 1 day of oocyte retrieval.
  vaginal, cervical and endometrial samples will be compared at the time of oocyte retrieval.

SECONDARY OUTCOMES:
Next generation sequencing techniques and qPCR will be used to assess the microbiota.I.e. measure of relative abundances and absolute abundances | This outcome data is measured at the 1 day of oocyte retrieval.
  qPCR to assess the microbiota. I.e. a quantitative measure Copies/mL. 16S V4 to investigate relative abundances

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Bernabeu, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided
WE plan to share all information allowed as per national law.